CLINICAL TRIAL: NCT01539837
Title: A Pilot Clinical Trial With the Iron Chelator Deferiprone in Parkinson's Disease
Acronym: DeferipronPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICL-11/SC/0101; 2011-001148-31 (EudraCT Number); 11/SC/0101 (Other: Research Ethics Committee)
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Brain Iron; Iron chelation; Oxidative stress
MeSH Terms: conditions — Parkinson Disease | interventions — Deferiprone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Drug excipient
  Interventions: Drug: Placebo
- Deferiprone 20mg (Active Comparator): 20mg/kg/day deferiprone
  Interventions: Drug: Deferiprone 20mg
- Deferiprone 30mg (Active Comparator): 30mg/kg/day Deferiprone
  Interventions: Drug: Deferiprone 30mg

INTERVENTIONS:
Drug: Deferiprone 20mg — 20mg/kg/d Deferiprone divided into two equal doses (morning and evening), every day for 6 months
  Other Names: Ferriprox
  Arms: Deferiprone 20mg
Drug: Placebo — Feriprox placebo administered orally at the same dosing volume as the 20mg/kg/day feriprox per day
  Other Names: Feriprox placebo
  Arms: Placebo
Drug: Deferiprone 30mg — 30mg/kg/d Deferiprone divided into two equal doses (morning and evening), every day for 6 months
  Other Names: Ferriprox
  Arms: Deferiprone 30mg

SUMMARY:
Parkinson's disease (PD) is a common neurodegenerative disease affecting movement. Although drug treatments for PD are available they only treat the symptoms of the disease, fail to halt neuronal loss, and are associated with long term side effects and loss of efficacy. There is a chronic need to develop neuroprotective therapies. Increased iron and oxidative stress have been heavily implicated in the neurodegenerative process in PD, hence removal of excess iron by iron chelation represents a potential drug target. Iron chelators are extensively utilised to treat peripheral iron overload disorders (e.g. thalassaemia) and recently the investigators have demonstrated iron chelators such as Deferiprone can enter the brain removing excess iron and are neuroprotective in PD animal models. Although good tolerability and efficacy to remove brain iron has also been shown in a pilot study with the iron chelators Deferiprone in young patients with Friedreich Ataxia, where iron accumulates in the dentate nucleus, no studies have been conducted in aged individuals affected by PD. Hence the aims of this study are 1) to assess whether Deferiprone is well tolerated in PD patients, 2) whether Deferiprone can remove the excess iron levels found in the brain area affected by PD, the substantia nigra, as assessed by Magnetic resonance imaging (MRI) and 3) whether Deferiprone has any direct effect on the clinical symptoms of PD. Three groups of 12 (total 36) early stage drug free PD patients will be treated with 20 or 30mg/kg/d Deferiprone or Placebo for 6 months. Over the 6 months patients will receive serial MRI scans, neurological examinations not only to assess PD symptoms but also psychological state, plus blood test to monitor for potential side effects. Positive results from this pilot will help support larger clinical trials to evaluate whether Deferiprone can slow down/halt PD.

DETAILED DESCRIPTION:
BACKGROUND Parkinson's disease (PD) is a progressive neurodegenerative disorder that affects approximately 2% of the population aged over 60 years. The common clinical motor control features are tremor, bradykinesia, postural abnormality and rigidity. However, in many patients non-motor features such as cognitive decline, depression, autonomic disturbances also occur as the disease progresses. The principal pathology is the degeneration of the nigrostriatal dopaminergic system which plays a major role in movement control through the release of dopamine in the striatum. Current therapeutic approach focus on dopamine replacement strategies either through the dopamine precursor L-DOPA or the use of dopamine agonists, and/or the use of monoamine oxidase inhibitors or catecholamine transferase inhibitors which prevent the breakdown of dopamine or facilitate L-DOPA entry into the brain. However, such therapeutic approaches are associated with declining efficacy and long term complications e.g. dyskinesias. Additionally, such therapeutic approaches only treat the clinical symptoms of PD and due not protect the neurons against degeneration hence the disease continues to progress with the patient experiencing increasing disability. Hence there is a chronic need for the development of neuroprotective drugs which prevent further neuronal loss and thus prevent the progression of the disease.

RATIONALE FOR CURRENT STUDY Hypothesis: Increased iron and oxidative stress play a major role in the neurodegenerative process in PD and iron chelation therapy can be effective in removing excess iron from the brain and potentially slowing the neurodegenerative process.

Research question: Can iron chelation therapy with Deferiprone remove excess iron in the substantia nigra in PD patients without toxic side effects. What effect does Deferiprone therapy have on the severity of PD and other brain function e.g. cognition, depression etc.

Increased iron levels have been heavily implicated in the neurodegenerative process in PD. Although many of our cellular processes require iron, when in excessive amounts it can trigger the formation of toxic chemicals called free radicals, of which there is extensive evidence of their increased formation in the PD brain. Hence removal of excess iron by iron chelation (drugs which bind and detoxify iron) represents a potential drug target.

Iron chelators e.g. Deferiprone in doses around 100mg/kg/day, are extensively utilised to treat peripheral iron overload disorders such as beta thalassaemia, where the patients requires regular blood transfusions but iron accumulates in the body when the red blood cells are removed from the circulation. Iron chelation therapy in such patients is associated with minimal side effects with long term use. Recently, in animal models of brain iron overload, we have demonstrated iron chelators can enter the brain removing excess iron. Additionally, we have recently shown that iron chelation therapy protects neurons against toxins in animal models of PD.

In 2007 20 or 30mg/kg/day Deferiprone was used in a pilot clinical trial in Friedreich ataxia (FA)patients, to assess whether the drug was well tolerated, removed excess brain iron and improved the clinical symptoms of FA. FA occurs due to a gene defect leading iron accumulation in the mitochondria in the cerebellum, toxicity of which leads to ataxia or inability to control muscle movements. FA is diagnosed in young individuals (14-26 years of age) and has no clinical treatment. In this 6 months FA study Deferiprone at 20 or 30mg/kg/day was well tolerated by the patients and resulted in a reduction in brain iron, as indicated by MRI brain imaging, and led to a clinical improvement in patient symptoms. Whilst this represents the first clinical use of an iron chelator to treat a neurodegenerative disorder, the FA patients in this study were young (14-23 years old) hence we do not know how aged (average age 60years) individuals commonly affected by PD will respond to iron chelator treatment. Hence the first aim of this study is to conduct the first pilot clinical trial with an iron chelator in newly diagnosed PD patients to assess tolerability along with its ability to reduce iron content in the brain area affected in PD, the substantia nigra, as assessed by MRI.

A number of clinical trials have already been conducted in PD with potential neuroprotective drugs but their ability to slow the disease process has been controversial since these drugs have a direct effects on the symptoms of PD itself. Hence it is difficult to say whether the beneficial effects of the drugs are due the prevention of further neuronal loss thus slowing the disease or whether they improve the patient's ability to move directly. PD progresses in most patients fairly slowly, hence we don't expect to see detectable neuroprotection following 6 months Deferiprone treatment but it will allow us to assess whether Deferiprone therapy has any direct effects on PD symptoms. Hence the second aim of this study will be to examine whether iron chelation therapy has a direct effect on PD symptomology.

If this pilot study clearly demonstrates good tolerability of Deferiprone in PD patients whilst showing good removal of excess SN iron level yet having minimal direct effect on PD symptomology this data will form the basis of large funding application for a multicentre clinical trials to investigate whether long term Deferiprone treatment can slow/halt the progression of PD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease
* disease duration less than 5 years
* stable response to standard anti-Parkinson's medication for at least 6 weeks

Exclusion Criteria:

* Other neurological conditions
* Diabetes
* Renal or liver disease
* Blood disorders
* Pregnancy or breast feeding
* Conditions which cause immunocompromise e.g. episodes of neutropaenia or agranulocytosis, HIV etc
* Prior history of hypersensitivity to Deferiprone or its excipient
* Pacemaker
* artificial heart valves
* ever had surgery to the head
* Metalic implants in the CNS e.g. cerebral aneurysm clips
* history of metal entering the eye

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David T Dexter, PhD, Principal Investigator — Imperial College London
Locations (1):
- Centre for Neuroscience, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dexter DT, Wells FR, Agid F, Agid Y, Lees AJ, Jenner P, Marsden CD. Increased nigral iron content in postmortem parkinsonian brain. Lancet. 1987 Nov 21;2(8569):1219-20. doi: 10.1016/s0140-6736(87)91361-4. No abstract available. PMID 2890848
- [Background] Oakley AE, Collingwood JF, Dobson J, Love G, Perrott HR, Edwardson JA, Elstner M, Morris CM. Individual dopaminergic neurons show raised iron levels in Parkinson disease. Neurology. 2007 May 22;68(21):1820-5. doi: 10.1212/01.wnl.0000262033.01945.9a. PMID 17515544
- [Background] Ward RJ, Dexter D, Florence A, Aouad F, Hider R, Jenner P, Crichton RR. Brain iron in the ferrocene-loaded rat: its chelation and influence on dopamine metabolism. Biochem Pharmacol. 1995 Jun 16;49(12):1821-6. doi: 10.1016/0006-2952(94)00521-m. PMID 7598744
- [Background] Dexter DT, Statton SA, Whitmore C, Freinbichler W, Weinberger P, Tipton KF, Della Corte L, Ward RJ, Crichton RR. Clinically available iron chelators induce neuroprotection in the 6-OHDA model of Parkinson's disease after peripheral administration. J Neural Transm (Vienna). 2011 Feb;118(2):223-31. doi: 10.1007/s00702-010-0531-3. Epub 2010 Dec 17. PMID 21165659
- [Background] Boddaert N, Le Quan Sang KH, Rotig A, Leroy-Willig A, Gallet S, Brunelle F, Sidi D, Thalabard JC, Munnich A, Cabantchik ZI. Selective iron chelation in Friedreich ataxia: biologic and clinical implications. Blood. 2007 Jul 1;110(1):401-8. doi: 10.1182/blood-2006-12-065433. Epub 2007 Mar 22. PMID 17379741
- [Result] Martin-Bastida A, Ward RJ, Newbould R, Piccini P, Sharp D, Kabba C, Patel MC, Spino M, Connelly J, Tricta F, Crichton RR, Dexter DT. Brain iron chelation by deferiprone in a phase 2 randomised double-blinded placebo controlled clinical trial in Parkinson's disease. Sci Rep. 2017 May 3;7(1):1398. doi: 10.1038/s41598-017-01402-2. PMID 28469157

RESULTS

PARTICIPANT FLOW:
Groups:
- Deferiprone 20mg: 20mg/kg/day deferiprone divided into two equal doses (morning and evening), every day for 6 months
- Deferiprone 30mg: 30mg/kg/day Deferiprone divided into two equal doses (morning and evening), every day for 6 months
Period: Overall Study
Arm/Group | Placebo | Deferiprone 20mg | Deferiprone 30mg
Started | 8 | 7 | 7
Completed | 8 | 6 | 5
Not Completed | 0 | 1 | 2
Not completed — reduce neutrophil level | 0 | 1 | 1
Not completed — bad compliance | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Deferiprone 20mg | Deferiprone 30mg | Total
Number analyzed (Participants) | 8 | 7 | 7 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.38 (3.23) | 68.57 (2.17) | 62.85 (2.74) | 65.26 (2.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 2 | 10
  Male | 3 | 4 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 7 | 7 | 22
Parkinson's disease duration [Mean (Standard Deviation); unit: years] | 3.54 (0.34) | 2.82 (0.69) | 3.02 (2.69) | 3.12 (1.24)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events
Description: To assess whether there were any serious adverse events in 6-month treatment with Deferiprone.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Deferiprone 20mg | Deferiprone 30mg
Number analyzed (Participants) | 8 | 7 | 7
Participants | 0 | 0 | 0

2. Secondary Outcome: Iron Concentrations in the Dentate Nucleus
Description: Assess whether Deferiprone therapy directly affects the symptoms of Parkinson's disease, modify regional brain mineralization (iron concentration) as assessed with T2* MRI in PD patients in the dentate nucleus. In previous animal studies, Deferiprone treatment reduced dentate nucleus iron content, as assessed by MRI. An increase in the T2*MRI value represents an increase in mineralization.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: ms
Arm/Group | Placebo | Deferiprone 20mg | Deferiprone 30mg
Number analyzed (Participants) | 8 | 7 | 7
ms | 30.74 (0.65) | 30.59 (0.87) | 29.86 (1.10)
Statistical Analysis 1: Comparison: Placebo vs Deferiprone 20mg vs Deferiprone 30mg; Test type: Superiority; p < 0.01, Pairwise comparisons,post-hoc Bonferoni — calculated

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Placebo | Deferiprone 20mg | Deferiprone 30mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 6/7 | 6/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | Deferiprone 20mg (N=7) | Deferiprone 30mg (N=7)
Decline in white cell counts (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal upset (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Muscular joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes